CLINICAL TRIAL: NCT06475989
Title: A Randomized Phase III Study of BRAF-Targeted Therapy vs Cabozantinib in RAI-Refractory Differentiated Thyroid Cancer With BRAF V600Em
Brief Title: Study of Targeted Therapy vs. Chemotherapy in Patients With Thyroid Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA3231; NCI-2024-03023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA3231 (Other: ECOG-ACRIN Cancer Research Group); EA3231 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-17; First posted 2024-06-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Refractory Differentiated Thyroid Gland Carcinoma
MeSH Terms: interventions — Specimen Handling; cabozantinib; dabrafenib; Magnetic Resonance Spectroscopy; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Dabrafenib and trametinib) (Active Comparator): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Drug: Trametinib
- Arm B (Cabozantinib) (Experimental): Patients receive cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, blood sample collection and may undergo MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib — Given PO
  Arms: Arm B (Cabozantinib)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
  Arms: Arm A (Dabrafenib and trametinib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary study
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK-1120212; GSK1120212; JTP-74057; MEK Inhibitor GSK1120212
  Arms: Arm A (Dabrafenib and trametinib)

SUMMARY:
This phase III trial compares the effect of cabozantinib versus combination dabrafenib and trametinib for the treatment of patients with differentiated thyroid cancer that does not respond to treatment (refractory) and which expresses a BRAF V600E mutation. Cabozantinib is in a class of medications called receptor tyrosine kinase inhibitors. It binds to and blocks the action of several enzymes which are often over-expressed in a variety of tumor cell types. This may help stop or slow the growth of tumor cells and blood vessels the tumor needs to survive. Dabrafenib is an enzyme inhibitor that binds to and inhibits the activity of a protein called B-raf, which may inhibit the proliferation of tumor cells which contain a mutated BRAF gene. Trametinib is also an enzyme inhibitor. It binds to and inhibits the activity of proteins called MEK 1 and 2, which play a key role in activating pathways that regulate cell growth. This may inhibit the growth of tumor cells mediated by these pathways. The usual approach for patients with thyroid cancer is targeted therapy with dabrafenib and trametinib. This trial may help researchers decide which treatment option (cabozantinib alone or dabrafenib in combination with trametinib) is safer and/or more effective in treating patients with refractory BRAF V600E-mutated differentiated thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) in patients with BRAF V600Em differentiated thyroid cancer who progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

SECONDARY OBJECTIVES:

I. To compare the objective response rate in patients with BRAF V600Em differentiated thyroid cancer that progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

II. To compare the duration of response in patients with BRAF V600Em differentiated thyroid cancer that progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

III. To compare the overall survival in patients with BRAF V600Em differentiated thyroid cancer that progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

IV. To compare the PFS2 in patients with BRAF V600Em differentiated thyroid cancer that progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

V. To compare the safety/tolerability in patients with BRAF V600Em differentiated thyroid cancer that progressed on frontline multikinase inhibitor treated with dabrafenib/trametinib or cabozantinib.

QUALITY OF LIFE OBJECTIVE:

I. To assess patient tolerability of treatment using the Functional Assessment Cancer Therapy General (FACT G)P5 and general quality of life using the FACT-G7.

OUTLINE: Patients are randomized to 1 of 2 arms. Patients may crossover to other treatment arm at the time of progression.

ARM A: Patients receive dabrafenib orally (PO) twice per day (BID) and trametinib PO once per day (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, blood sample collection and may undergo magnetic resonance imaging (MRI) throughout the study.

ARM B: Patients receive cabozantinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, blood sample collection and may undergo MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient must have differentiated thyroid cancer (DTC) with BRAF V600E mutation as determined by local testing, including the following subtypes (Note: results of a previous biopsy will be accepted):

  * Papillary thyroid carcinoma including histological variants of papillary thyroid carcinoma (PTC) such as follicular variant, tall cell, columnar cell, cribriform-morular, solid, oxyphil, Warthin-like, trabecular, tumor with nodular fasciitis-like stroma, Hürthle cell variant of papillary carcinoma, poorly differentiated.
  * Follicular thyroid carcinoma including histological variants of follicular thyroid carcinoma (FTC) such as Hürthle cell, clear cell, insular, and poorly differentiated
* Patient must have been previously treated with or deemed ineligible for treatment with Iodine-131 for DTC, and must be receiving thyroxine suppression therapy
* Patient must have had prior treatment with at least one of the following vascular endothelial growth factor receptors (VEGFR)-targeting tyrosine kinase inhibitor (TKI) agents for DTC: lenvatinib or sorafenib.

  * NOTE: Up to two prior VEGFR-targeting TKI agents are allowed including, but not limited to lenvatinib and sorafenib
* Patient must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1·1 on chest CT (computed tomography)/abdominal/pelvis CT/MRI (magnetic resonance imaging) performed within 4 weeks prior to randomization
* Patient must have radiographic progression by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 over any time interval on or after most recent prior systemic treatment
* Patient must not have any of the following cardiovascular and thromboembolic disorders or medical conditions:

  * Congestive heart failure class 3 or 4 as defined by the New York Heart Association, unstable angina pectoris, or serious cardiac arrhythmias.
  * Uncontrolled hypertension defined as sustained blood pressure > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
  * Stroke, myocardial infarction, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months prior to randomization. Patients with more recent diagnosis of deep venous thrombosis are allowed if stable and treated with therapeutic anticoagulation for at least 6 weeks prior to randomization
* Patient must not have any clinically significant hematemesis or haemoptysis of > 0·5 teaspoon (> 2·5 mL) of red blood or history of other significant bleeding within 3 months prior to randomization
* Patient must not have any cavitating pulmonary lesion(s) or lesions invading major pulmonary blood vessels
* Patient must not be on any concomitant anticoagulation with oral anticoagulants or platelet inhibitors, except for the following allowed agents:

  * Low-dose aspirin for cardioprotection.
  * Therapeutic anticoagulation with any agent in patients (1) without known brain metastases, (2) on a stable dose for at least 6 weeks prior to randomization, and (3) with no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Patient must not have any gastrointestinal (GI) disorders associated with a high risk of perforation or fistula formation:

  * Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction
  * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months prior to randomization
* Patient must have completed any prior local therapy (e.g., surgery, radiation, ablation) at least 4 weeks prior to randomization, with complete wound healing and resolution of clinically relevant complications from prior local therapy
* Patient must not have had major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to randomization. Complete wound healing from major surgery must have occurred 4 weeks prior to randomization and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days prior to randomization
* Patient must not have any lesion(s) with ≥ 2cm growth within 3 months or ≥ 1.5cm growth within 2 months prior to randomization, and must not have documented anaplastic histology at or following cancer recurrence
* Patient must not have had prior treatment with cabozantinib or any prior BRAF targeted therapy for thyroid cancer
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.

A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

* Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 2 weeks after the last dose of dabrafenib and 4 months after the last dose of trametinib or cabozantinib. Patients must also not breastfeed while on study treatment and for 2 weeks after the last dose of dabrafenib and for 4 months after the last dose of trametinib or cabozantinib.

  * NOTE: Patients of childbearing potential who are on hormonal contraceptives may be at risks because dabrafenib may decrease the efficacy of hormonal contraceptives. An effective non-hormonal contraception should be used during therapy and for 2 weeks following discontinuation of dabrafenib and at least 4 months following the last dose of trametinib and cabozantinib
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Hemoglobulin (Hgb) ≥ 8 g/dL obtained ≤ 28 days prior to protocol randomization
* Leukocytes ≥ 3,000/mcL obtained ≤ 28 days prior to protocol randomization
* Absolute neutrophil count (ANC) ≥ 1,500/mcL obtained ≤ 28 days prior to protocol randomization
* Platelets ≥ 100,000/mcL obtained ≤ 28 days prior to protocol randomization
* Total bilirubin ≤ 2.0 x institutional upper limit of normal (ULN) obtained ≤ 28 days prior to protocol randomization
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 × institutional ULN or < 5.0 x ULN with the presence of hepatic metastasis obtained ≤ 28 days prior to protocol randomization
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m² obtained ≤ 28 days prior to protocol randomization
* Urine protein/creatinine (UPC) ratio ≥ 1 obtained ≤ 28 days prior to protocol randomization
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging obtained after central nervous system (CNS)-directed therapy (radiotherapy and/or surgery) shows no evidence of progression. CNS disease must be stable for at least 4 weeks prior to randomization; patients must be neurologically asymptomatic and without corticosteroid treatment at time of randomization
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients must have corrected QT interval calculated by the Fridericia formula (QTcF) ≤ 500 ms obtained within 28 days prior to randomization.

  * NOTE: If a single electrocardiogram (ECG) shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 minutes (min) must be performed within 30 min after the initial ECG, and the average of these 3 consecutive results for QTcF will be used to determine eligibility
* Patient must be English or Spanish speaking to be eligible for the quality of life (QOL) component of the study.

  * NOTE: Sites cannot translate the associated QOL forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to radiographic progression of disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death from any cause, up to 5 years
  PFS will be compared between the two groups using a stratified log-rank test with one-sided type I error of 0.05. Median PFS and 95% confidence interval (CI) for each treatment arm will be estimated using the Kaplan-Meier method. The stratified hazard ratio and 95% CI will be estimated using a Cox proportional hazard model with treatment group as the independent variable.

SECONDARY OUTCOMES:
Objective response | Up to 5 years
  Will be assessed based on international criteria proposed by the RECIST 1.1 guideline. Response (complete and partial responses) rate will be estimated. Will be compared using the Fisher's exact test.
Overall survival | From randomization to death from any cause, up to 5 years
  Median and 95% CI will be estimated in each arm using the Kaplan-Meier method.
Duration of response | From confirmed response (complete response or partial response) to progression among patients who achieve a response, up to 5 years
  Median and 95% CI will be estimated in each arm using the Kaplan-Meier method.
PFS2 - the time from randomization to progression on subsequent therapy or death from any cause (whichever occurs first) | From randomization to progression on subsequent therapy or death from any cause, up to 5 years
  Median and 95% CI will be estimated in each arm using the Kaplan-Meier method. PFS2 will be measured for every patient. For patients who receive a next line of therapy, PFS2 will be measured from the time of randomization to radiographic progression on the next line of therapy after the protocol-assigned therapy, or death from any cause, whichever occurs first. If patients are alive and have not had progression on the next of line therapy, they will be censored at the last assessment on the next line of therapy, and PFS2 will be measured from the time of randomization to the last assessment. For patients who do not receive the next line of therapy, PFS2 will be measured from the time of randomization to last assessed on the protocol-assigned therapy and will be censored unless death occurs, in which case death will count as an event.
Incidence of adverse events | at 2 weeks, 4 weeks, 8 weeks, 16 weeks, and then every 12 weeks after the 16-week confirmatory scan
  Using the National Cancer Institute's Common Terminology Criteria for Adverse Events. Response rate and grade 3 or higher toxicity rates will be compared using the Fisher's exact test between the two arms.

OTHER OUTCOMES:
Patient tolerability | At baseline, 4, 8, 16, and 28 weeks
  Will assess patients tolerability of treatment using the Functional Assessment of Cancer Therapy-General (FACT G)7.

CONTACTS AND LOCATIONS:
Overall Officials: Lova Sun, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (112):
- United States (112):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming